CLINICAL TRIAL: NCT04430244
Title: Deep Anterior Lamellar Keratoplasty Using Dehydrated Versus Standard Organ Culture Stored Donor Corneas: A Randomized Controlled Trial
Brief Title: Deep Anterior Lamellar Keratoplasty Using Dehydrated Versus Standard Organ Culture Stored Donor Corneas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Internazionale di Ricerca e Formazione in Oftalmologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020001
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DALK using Dehydrated Corneas (Experimental): Corneal transplantation of anterior lamellar grafts from dehydrated corneas.
  Interventions: Procedure: Deep anterior lamellar keratoplasty
- DALK using Standard Organ Culture Stored Corneas (Active Comparator): Corneal transplantation of anterior lamellar grafts from standard organ culture stored corneas.
  Interventions: Procedure: Deep anterior lamellar keratoplasty

INTERVENTIONS:
Procedure: Deep anterior lamellar keratoplasty — Deep anterior lamellar keratoplasty using dehydrated corneas
  Arms: DALK using Dehydrated Corneas
Procedure: Deep anterior lamellar keratoplasty — Deep anterior lamellar keratoplasty using standard organ culture stored corneas
  Arms: DALK using Standard Organ Culture Stored Corneas

SUMMARY:
The objective of this study is to assess the outcomes between deep anterior lamellar keratoplasty using dehydrated versus standard organ culture stored donor corneas.

DETAILED DESCRIPTION:
Keratoconus is a common corneal disease characterized by progressive thinning and steepening resulting in significant visual impairment. With improved instrumentation and corneal imaging technology, deep anterior keratoplasty has been recognized as the preferred primary operative technique for cases of keratoconus requiring corneal transplantation.

Since corneas preserved through organ culture remain viable only for up to 4 weeks, techniques that can extend storage of corneas have been explored.

The objective of this study is to assess the outcomes between deep anterior lamellar keratoplasty using dehydrated versus standard organ culture stored donor corneas.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus
* Surgical candidates for deep anterior lamellar keratoplasty

Exclusion Criteria:

* Ocular comorbidities other than cataract (ie. visual significant optic nerve or macular disease)
* Previous corneal transplantations or other ocular surgeries except uncomplicated cataract surgery
* Inability to comply with study protocol or participate in follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in best spectacle-corrected visual acuity | Preoperatively; and 6 and 12 months postoperatively
  Measured as the difference in best spectacle-corrected visual acuity preoperative, 6 and 12 months postoperatively using ETDRS chart

SECONDARY OUTCOMES:
Change in astigmatism | Preoperatively; and 6 and 12 months postoperatively
  Topographic astigmatism (Diopters) is measured using anterior segment optical coherence tomography (CASIA)
Change in Thinnest-point pachymetry | Preoperatively; and 6 and 12 months postoperatively
  Thinnest-point pachymetry values (um) are measured using anterior segment optical coherence tomography (CASIA)
Change in endothelial cell density | Preoperatively; and 6 and 12 months postoperatively
  Measured using noncontact specular microscopy
Incidence of graft rejection | 6 and 12 months postoperatively
  Clinically assessed during postoperative examinations
Incidence of graft failure | 6 and 12 months postoperatively
  Clinically assessed during postoperative examinations
Corneal donor loss due to preparation | Intraoperative
  Based on intraoperative assessment of corneas unusable for corneal transplantation

OTHER OUTCOMES:
Refraction | 6 and 12 months postoperatively
  Measured by manifest refraction
Adverse Events/Complication | up to 12 months postoperatively
  Comparison of total rates of adverse events/complications assessed clinically

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Busin, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Ospedali Privati Forlì "Villa Igea", Forlì, Emilia-Romagna, Italy